CLINICAL TRIAL: NCT03617315
Title: Crosslinked Hyaluronic Acid With Liposomes and Crocin in the Treatment of Dry Eye Disease Due to Moderate Meibomian Glands Dysfunction
Brief Title: Crosslinked Hyaluronic Acid With Liposomes and Crocin in Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, José-María Sánchez-González, PhD Optometry and Vision Science, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HyaluronicAcidClinicalTrial
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction; Dry Eye Syndromes
Keywords: Crosslinked Hyaluronic Acid; Meibomian Gland Disfunction; Lubricants; Contact Lens; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — poly(vinyl alcohol)-hylauronic acid

STUDY DESIGN:
Intervention Model Description: Contralateral Eye Study
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients did not know the artificial tear that should be applied. The researcher in charge of processing the results and drawing the conclusions did not know the name of the artificial tears
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid (Experimental): One drop application of Hyaluronic acid + Galact-Xyloglucan with a dosage of 3 times a day for 45 days
  Interventions: Drug: Hylauronic Acid
- CrossLinked Hyalurnic Acid (Experimental): One drop application of Crosslinked Hylauronic Acid + Liposomes with a dosage of 3 times a day for 45 days
  Interventions: Drug: Hylauronic Acid

INTERVENTIONS:
Drug: Hylauronic Acid — Schirmer Test, BUT test and OSDI test. Previous and After treatment
  Other Names: Galacto-Xiloglucan; HA+GX

SUMMARY:
A total of 50 eyes were analyzed (25 patients). The subjects selected were over 18 years of age. No gender distinction was made in the choice of subjects. All subjects were carriers of silicone hydrogel contact lenses. The antecedents of the eye diseases not identified, neither the previous eye surgeries nor the systemic or ocular medication. All patients read, understood and signed an informed consent form of the study.

DETAILED DESCRIPTION:
A study was performed using the contralateral eye, the study groups were randomized. The choice of eye for each tear was random and established as an artificial tear A and artificial tear B. The patients were not previously warned about the type of artificial tear they were going to use or the difference that existed between them, therefore, they were unaware of the benefits that such tears could offer them. The examiner did know what tear was applied to each eye.

As for the lubricants used; Tear A (Aquoral Forte®, ESTEVE®, Farmigea, Pisa, Italy) was a combination of 0.4% unridged hyaluronic acid and 0.2% Galacto-xyloglucan. The galacto-xyloglucan is extracted from the tamarind seed. It consists of 30 single doses, each with 0.5 ml and have a daily use closure, that is, it can not be used once 12 hours have passed since the dose was opened. This lubricant lacks preservatives.

On the other hand, tear B (Aquoral Lipo® [Spain] / Lumixa® [Italy], ESTEVE®, Farmigea, Pisa, Italy) is a combination of three components; cross-linked hyaluronic acid (CXL) at 0.15%, crocin and liposomes. It is an ophthalmic lubricant and antioxidant solution. Its package is 10 ml multidose, so it can be used for a long time. It is composed of liposomes, sodium salt of crosslinked hyaluronic acid 0.15%, ethylenediaminetetraacetic acid (EDTA) disodium salt and crocin. Although this tear comes in a multi-dose container, it does not contain a preservative due to the dispenser that does not let microorganisms from outside. Contact lenses can be used while both lubricants are applied. In this regard, the study patients used their silicone hydrogel contact lenses monthly during the study.

All patients in the study had a period of one month without using any type of artificial tear or eye drops. Once this time or study was over, the patients were explained how artificial tears should be instilled. The visits were carried out blindly by research optometrists. Who did not know how the distribution of artificial tears in patients had been. The artificial tears were administered 3 times a day for 6 weeks and the subjects belonging to the study underwent a clinical examination in the period prior to treatment and 45 days after the treatment, once the treatment with artificial tears. He was repeated the tests of the beginning, nevertheless, the meibografía was not realized, since the use of artificial tears was not going to cause the growth of the glands of Meibomio

ELIGIBILITY:
Inclusion Criteria:

* Ocular Surface Disease Index over 15
* Dysfunction of the meibomian gland
* User contact lenses silicone hydrogel
* User of digital screens for a long timeç

Exclusion Criteria:

* Previous eye surgeries
* Previous eye pathologies
* User of artificial tears
* User of ophthalmic gels

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Schirmer Test | 6 weeks
  Measurement of the tear volume. Scale between 0 and 30 milimeters (mm) Higger is better
Break Up Time Test | 6 weeks
  Lacrimal rupture time of the lipid layer. Scale between 0 and 25 seconds (s) Higger is better
Ocular Surface Disease Index | 6 weeks
  Dry Eye Score from Questionnaire. Scale between 0 and 50 points. Higger is worse

CONTACTS AND LOCATIONS:
Locations (1):
- José-María Sánchez-González, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
Share with University of Seville Researches through the virtual learning platform

REFERENCES:
- [Result] Fallacara A, Vertuani S, Panozzo G, Pecorelli A, Valacchi G, Manfredini S. Novel Artificial Tears Containing Cross-Linked Hyaluronic Acid: An In Vitro Re-Epithelialization Study. Molecules. 2017 Nov 30;22(12):2104. doi: 10.3390/molecules22122104. PMID 29189737
- [Result] Uccello-Barretta G, Balzano F, Vanni L, Sanso M. Mucoadhesive properties of tamarind-seed polysaccharide/hyaluronic acid mixtures: A nuclear magnetic resonance spectroscopy investigation. Carbohydr Polym. 2013 Jan 16;91(2):568-72. doi: 10.1016/j.carbpol.2012.07.085. Epub 2012 Aug 25. PMID 23121946
- [Result] Doan S, Bremond-Gignac D, Chiambaretta F. Comparison of the effect of a hyaluronate-trehalose solution to hyaluronate alone on Ocular Surface Disease Index in patients with moderate to severe dry eye disease. Curr Med Res Opin. 2018 Aug;34(8):1373-1376. doi: 10.1080/03007995.2018.1434496. Epub 2018 Feb 7. PMID 29381080
- [Result] Jacobi C, Kruse FE, Cursiefen C. Prospective, randomized, controlled comparison of SYSTANE UD eye drops versus VISINE INTENSIV 1% EDO eye drops for the treatment of moderate dry eye. J Ocul Pharmacol Ther. 2012 Dec;28(6):598-603. doi: 10.1089/jop.2012.0066. Epub 2012 Jul 19. PMID 22813209
- [Result] Postorino EI, Rania L, Aragona E, Mannucci C, Alibrandi A, Calapai G, Puzzolo D, Aragona P. Efficacy of eyedrops containing cross-linked hyaluronic acid and coenzyme Q10 in treating patients with mild to moderate dry eye. Eur J Ophthalmol. 2018 Jan;28(1):25-31. doi: 10.5301/ejo.5001011. Epub 2018 Feb 19. PMID 28777385
- [Result] Acar D, Molina-Martinez IT, Gomez-Ballesteros M, Guzman-Navarro M, Benitez-Del-Castillo JM, Herrero-Vanrell R. Novel liposome-based and in situ gelling artificial tear formulation for dry eye disease treatment. Cont Lens Anterior Eye. 2018 Feb;41(1):93-96. doi: 10.1016/j.clae.2017.11.004. Epub 2017 Dec 6. PMID 29223649
- [Result] Rolando M, Valente C. Establishing the tolerability and performance of tamarind seed polysaccharide (TSP) in treating dry eye syndrome: results of a clinical study. BMC Ophthalmol. 2007 Mar 29;7:5. doi: 10.1186/1471-2415-7-5. PMID 17394642
- [Result] Williams DL, Mann BK. Efficacy of a crosslinked hyaluronic acid-based hydrogel as a tear film supplement: a masked controlled study. PLoS One. 2014 Jun 10;9(6):e99766. doi: 10.1371/journal.pone.0099766. eCollection 2014. PMID 24914681